CLINICAL TRIAL: NCT02896647
Title: 3D Phase Sensitive Inversion Recuperation MRI to Detect and Characterize Multiple Sclerosis Spinal Cord Lesions
Acronym: ESPOIR
Status: Terminated | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2016_20
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
This study aims to assess the interest of 3D Phase Sensitive Inversion Recuperation (PSIR)sequence in the MRI detection of spinal cord lesion. It will compare the sensitivity of this MRI sequence compared to the T1 and T2 sequences recommended in the assessment of neuraxis inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* patients scheduled for spinal cord MRI exploration for the assessment of neuraxis inflammatory diseases

Exclusion Criteria:

* contraindication to MRI
* allergy to contrast media
* patient under legal protection
* no health insurance coverage
* patient's refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for spinal cord MRI exploration for the assessment of a neuraxis inflammatory disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
number of spinal cord lesions | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Augustin LECLER, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation A De Rothschild, Paris, France